CLINICAL TRIAL: NCT01727700
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety and Efficacy of Fixed-Dose Once-daily Oral Aripiprazole in Children and Adolescents With Tourette's Disorder
Brief Title: Study Evaluating the Safety and Efficacy of Fixed-dose Once-daily Oral Aripiprazole in Children and Adolescents With Tourette's Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31-12-293
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Results first posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Tourette's Disorder; Tic Disorder
Keywords: Tourette Syndrome; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Tic Disorders; Tics; Movement Disorders; Mental Disorders; Aripiprazole
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Tics; Movement Disorders; Mental Disorders | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Matching Placebo Once-Daily
  Interventions: Drug: Placebo
- Aripiprazole 5 mg or 10 mg (Experimental): Aripiprazole 5 mg or 10 mg Immediate Release Once-Daily
  Interventions: Drug: Aripiprazole
- Aripiprazole 10 mg or 20 mg (Experimental): Aripiprazole 10 mg 20 mg Immediate Release Once-Daily
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Once-daily, tablet
  Other Names: Abilify
  Arms: Aripiprazole 10 mg or 20 mg; Aripiprazole 5 mg or 10 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The goal of the current trial is to determine efficacy and safety of Once-daily aripiprazole in reducing Total Tic Severity in children and adolescents with Tourette's Disorder.

DETAILED DESCRIPTION:
Tourette's Disorder is a neuropsychiatric condition that is characterized by the appearance of tics that can be simple or complex in nature. A tic is a sudden, rapid, recurrent, non-rhythmic, stereotyped motor movement or vocalization. There are a very limited number of medications approved for the treatment of Tourette's Disorder. The goal of the current trial is to obtain efficacy, safety, and tolerability data in a controlled condition of a Once-daily aripiprazole formulation in children and adolescents with Tourette's Disorder. The trial has an 8-week long double-blind treatment period after a pretreatment (screening/washout phase), and the subjects will be followed up for 1 month after the last treatment. The Once-daily tablet formulation that will be evaluated in this trial represents a daily dosage regimen that is intended to be administered to children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* male or female, 7 to 17 year old (inclusive) at the time of signing consent
* meets DSM-IV-TR diagnostic criteria for Tourette's Disorder
* Presenting tic symptoms cause impairment in the subject's normal routines, which include academic achievement, occupational functioning, social activities, and/or relationships
* Females of childbearing potential must have a negative pregnancy test, must be practicing acceptable double-barrier methods of contraception and must not be pregnant or lactating
* Written informed consent obtained from a legally acceptable representative & informed assent at Screening as applicable by trial center's IRB/IEC
* The subject, designated guardian(s) or caregiver(s) are able to comprehend and satisfactorily comply with the protocol requirements, as evaluated by the investigator

Exclusion Criteria:

* Clinical presentation and/or history, consistent with another neurologic condition that may have accompanying abnormal movements
* History of schizophrenia, bipolar disorder, or other psychotic disorder
* Subject receiving psychostimulants for treatment of ADD/ADHD and who have developed and/or had exacerbations of tic disorder after initiation of stimulant treatment
* Currently meets DSM-IV-TR criteria for a primary mood disorder
* Severe Obsessive Compulsive Disorder (OCD)
* Taken aripiprazole within 30 days of the Screening visit
* Received any investigational agent in a clinical trial within 30 days prior to Screening, enrolled in studies 31-12-272, 31-12-273, 31-12-274; or who were randomized into a clinical trial with Once-daily aripiprazole at any time
* History of neuroleptic malignant syndrome
* Sexually active patients not using 2 approved methods of contraception
* Females breastfeeding or pregnant (positive blood pregnancy test prior to receiving trial drug)
* Risk of committing suicide
* Body weight lower than 16 kg
* Taken neuroleptic or antiparkinson drugs < 14 days prior to randomization
* Requiring cognitive behavioral therapy (CBT) for Tourette's during trial
* Subject meets DSM-IV-TR criteria for any significant psychoactive substance use disorder within the past 3 months
* Positive drug screen
* Subject requires medications not allowed per protocol
* Use of CYP2D6 and CYP3A4 inhibitors or CYP3A4 inducers within 14 days prior to dosing and for duration of trial
* Use of herbal medications of any kind and nutritional or dietary supplements for Tourette's disorder within 7 days prior to dosing and for the duration of the trial
* Inability to swallow tablets or tolerate oral medication
* Abnormal laboratory test results, vital signs and ECG results

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kohegyi, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (75):
- United States (55):
  - Dothan, Alabama
  - Goodyear, Arizona
  - Tucson, Arizona
  - Corona, California
  - Sacramento, California
  - San Diego, California
  - Santa Ana, California
  - Wildomar, California
  - Norwich, Connecticut
  - Bradenton, Florida
  - Gainsville, Florida
  - Leesburg, Florida
  - Maitland, Florida
  - Miami, Florida
  - Orange City, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Savannah, Georgia
  - Naperville, Illinois
  - Indianapolis, Indiana
  - Overland Park, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Waldorf, Maryland
  - Bloomfield Hills, Michigan
  - Mount Arlington, New Jersey
  - Summit, New Jersey
  - Albuquerque, New Mexico
  - Manhasset, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Philadelphia, Pennsylvania
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Orem, Utah
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Henrico, Virginia
  - Norfolk, Virginia
  - Bellevue, Washington
  - Bothell, Washington
  - Middleton, Wisconsin
- Canada (4):
  - Kentville, Nova Scotia
  - Parry Sound, Ontario
  - Toronto, Ontario
  - Whitby, Ontario
- Germany (4):
  - Dresden, Germany
  - Freiburg im Breisgau, Germany
  - Mannheim, Germany
  - Würzburg, Germany
- Hungary (2):
  - Budapest, Hungary
  - Szeged, Hungary
- Italy (3):
  - Catania, Italy
  - Milan, Italy
  - Roma, Italy
- Mexico (3):
  - Mexico City, Mexico City
  - Durango, Mexico
  - Leon, Mexico
- Romania (2):
  - Bucharest, Romania
  - Iași, Romania
- Madrid, Spain, Spain
- Gothenburg, Sweden, Sweden

REFERENCES:
- [Derived] Sallee F, Kohegyi E, Zhao J, McQuade R, Cox K, Sanchez R, van Beek A, Nyilas M, Carson W, Kurlan R. Randomized, Double-Blind, Placebo-Controlled Trial Demonstrates the Efficacy and Safety of Oral Aripiprazole for the Treatment of Tourette's Disorder in Children and Adolescents. J Child Adolesc Psychopharmacol. 2017 Nov;27(9):771-781. doi: 10.1089/cap.2016.0026. Epub 2017 Jul 7. PMID 28686474

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 3, multicenter, randomized, double-blind, placebo-controlled trial in children and adolescents (aged 7-17 years) with Tourette's disorder (TD). 171 participants were screened, of which 133 were randomized to treatment.
Pre-assignment Details: The trial consisted of a pretreatment phase and a treatment phase. Pretreatment phase consisted of a screening and washout (when applicable) period. This was followed by an 8-week treatment phase starting with the baseline visit (Day 0). Particpants were randomized 1:1:1 to aripiprazole high dose, aripiprazole low dose or placebo.
Groups:
- Aripiprazole Low Dose: For participants who weighed < 50 kg at baseline, low dose was 5 mg/day. For participants who weighed ≥ 50 kg at baseline, low dose was 10 mg/day. All participants randomized to aripiprazole began treatment at 2 mg/day, with the dose titrated to 5 mg/day after 2 days. The dose was titrated to achieve the randomized dose. All participants were to have reached their randomized dose by Week 3 (Day 21) and were to remain on that dose.
- Aripiprazole High Dose: For participants who weighed < 50 kg at baseline, high dose was 10 mg/day. For participants who weighed ≥ 50 kg at baseline, high dose was 20 mg/day. All participants randomized to aripiprazole began treatment at 2 mg/day, with the dose titrated to 5 mg/day after 2 days. The dose was then titrated weekly until the randomized dose was achieved. All participants were to have reached their randomized dose by Week 3 (Day 21) and were to remain on that dose.
- Placebo: Participants received matching placebo tablets in the same way as aripiprazole.
Period: Overall Study
Arm/Group | Aripiprazole Low Dose | Aripiprazole High Dose | Placebo
Started | 44 | 45 | 44
Completed | 42 | 35 | 42
Not Completed | 2 | 10 | 2
Not completed — Adverse Event | 0 | 7 | 1
Not completed — Particpant withdrew consent | 0 | 3 | 1
Not completed — Protocol Violation | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole Low Dose | Aripiprazole High Dose | Placebo | Total
Number analyzed (Participants) | 44 | 45 | 44 | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.1 (3.1) | 11.8 (2.8) | 11.6 (2.8) | 11.5 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 11 | 29
  Male | 36 | 35 | 33 | 104

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS).
Description: The YGTSS is a semi-structured clinical interview designed to measure current (time frame of the past 1 week) tic severity. This scale consists of a tic inventory, with 5 separate rating scales to rate the severity of symptoms, and an impairment ranking. Ratings are made along 5 different dimensions on a scale of 0 to 5 for motor and vocal tics each, including number, frequency, intensity, complexity, and interference. Summation of these 10 scores (ie, 0-50) provides a TTS that was the primary outcome measure in this trial. The YGTSS ranking of impairment score rated on a 50-point scale anchored from 0 (no impairment) to 50 (severe impairment) to assess impairment experienced in areas of self-esteem, family life, social acceptance, and school scores. This is a fully validated scale in adults and has become a standard instrument for the evaluation of the severity of TD in children.
Time Frame: Baseline to Week 8
Population: Intent-to-Treat (ITT) Population: All participants randomly assigned to the double-blind treatment. At Week 8, data were available for 42 participants in the low dose, 35 in the high dose and 42 in the placebo group.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole Low Dose | Aripiprazole High Dose | Placebo
Number analyzed (Participants) | 42 | 35 | 42
Units on a scale | -13.35 (1.59) | -16.94 (1.61) | -7.09 (1.55)
Statistical Analysis 1: Comparison: Aripiprazole Low Dose vs Placebo; Assuming 5% of participants may drop out of the trial without a postbaseline efficacy evaluation, a total of 126 participants were required to provide at least 80% power to detect a treatment difference of -5 (common standard deviation [SD] of 8.5) between at least 1 of 2 aripiprazole dose levels and placebo in the primary outcome; Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis — The Hochberg procedure was used to adjust for multiplicity; Treatment, week, treatment by week interaction, region, and weight group were fixed categorical effects; baseline value as a fixed covariate; Treatment difference = -6.26, 95% CI 2-sided [-10.18 to -2.34]
Statistical Analysis 2: Comparison: Aripiprazole High Dose vs Placebo; Assuming 5% of participants may drop out of the trial without a postbaseline efficacy evaluation, a total of 126 participants were required to provide at least 80% power to detect a treatment difference of -5 (common standard SD of 8.5) between at least 1 of 2 aripiprazole dose levels and placebo in the primary outcome; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — The Hochberg procedure was used to adjust for multiplicity; [statistical method as in outcome 1, analysis 1]; Treatment difference = -9.85, 95% CI 2-sided [-13.84 to -5.86]

2. Secondary Outcome: Change in Clinical Global Impressions Scale-Tourette's Syndrome (CGI-TS) Score at Week 8.
Description: To assess CGI-TS severity, the rater or physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" However, the evaluation of illness was limited to manifestations of TD only. Response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients. The change score was obtained from CGI-TS improvement scale assessment: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Week 8
Population: ITT Population: All participants randomly assigned to the double-blind treatment. At Week 8, data were available for 42 participants in the low dose, 35 in the high dose and 42 in the placebo group.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole Low Dose | Aripiprazole High Dose | Placebo
Number analyzed (Participants) | 42 | 35 | 42
Units on a scale | 2.12 (0.21) | 2.13 (0.21) | 3.15 (0.2)
Statistical Analysis 1: Comparison: Aripiprazole Low Dose vs Placebo; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — The Hochberg procedure was used to adjust for multiplicity; [statistical method as in outcome 1, analysis 1]; Treatment difference = -1.03, 95% CI 2-sided [-1.54 to -0.52]
Statistical Analysis 2: Comparison: Aripiprazole High Dose vs Placebo; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — The Hochberg procedure was used to adjust for multiplicity; [statistical method as in outcome 1, analysis 1]; Treatment difference = -1.02, 95% CI 2-sided [-1.54 to -0.49]

3. Secondary Outcome: Mean Change From Baseline to Endpoint (Week 8) in Total YGTSS Score
Description: The YGTSS consists of a tic inventory, with 5 separate rating scales to rate the severity of symptoms (on a scale of 0 to 5 for 5 different dimensions, including number, frequency, intensity, complexity, and interference) of motor and vocal tics, and an impairment ranking. The Total YGTSS score is the summation of the severity scores of motor and vocal tics and also the ranking of impairment (range of 0 to 100). A missing value of a YGTSS item scale could result in a missing Total YGTSS score. A reduction in Total YGTSS score from baseline represents an improvement in symptoms.
Time Frame: Baseline to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole Low Dose | Aripiprazole High Dose | Placebo
Number analyzed (Participants) | 42 | 35 | 42
Units on a scale | -26.69 (3.34) | -32.80 (3.39) | -13.43 (3.27)
Statistical Analysis 1: Comparison: Aripiprazole Low Dose vs Placebo; Test type: Superiority or Other; p = 0.0017, Mixed Models Analysis — Treatment, week, treatment by week interaction, region, and weight group were fixed categorical effects; baseline value as a fixed covariate; Treatment difference = -13.26, 95% CI 2-sided [-21.43 to -5.08]
Statistical Analysis 2: Comparison: Aripiprazole High Dose vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Treatment difference = -19.37, 95% CI 2-sided [-27.70 to -11.04]

4. Secondary Outcome: Mean Change From Baseline to Endpoint (Week 8) in CGI-TS Severity Score
Description: The CGI-TS Severity scale (range 0-7) is a single-item rating score, with higher scores representing greater severity or less improvement. A response of 0 (not assessed) is considered and handled as missing data.
Time Frame: Baseline to Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole Low Dose | Aripiprazole High Dose | Placebo
Number analyzed (Participants) | 42 | 35 | 42
Units on a scale | -1.35 (0.19) | -1.47 (0.19) | -0.55 (0.19)
Statistical Analysis 1: Comparison: Aripiprazole Low Dose vs Placebo; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Treatment difference = -0.80, 95% CI 2-sided [-1.27 to -0.33]
Statistical Analysis 2: Comparison: Aripiprazole High Dose vs Placebo; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; MMRM = -0.92, 95% CI 2-sided [-1.41 to -0.44]

5. Secondary Outcome: Response Rate
Description: Clinical response is defined as > 25% improvement from baseline to Week 8 in YGTSS TTS or a CGI-TS Change score of 1 [very much improved] or 2 [much improved] at Week 8. Response will be considered as missing only if both YGTSS TTS and CGI-TS change score are missing. As long as one of them is non-missing, response outcome will be determined based on the non-missing score.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: Percentage of Responders
Arm/Group | Aripiprazole Low Dose | Aripiprazole High Dose | Placebo
Number analyzed (Participants) | 42 | 35 | 42
Percentage of Responders | 73.8 | 88.6 | 54.8
Statistical Analysis 1: Comparison: Aripiprazole Low Dose vs Placebo; Test type: Superiority or Other; p = 0.0835, Cochran-Mantel-Haenszel — P-value derived from Cochran-Mantel-Haenszel (CMH) General Association Test adjusting for region and weight group; Response ratio > 1 favors aripiprazole; Response ratio = 1.36, 95% CI 2-sided [0.98 to 1.88]
Statistical Analysis 2: Comparison: Aripiprazole High Dose vs Placebo; Test type: Superiority or Other; p = 0.0014, Cochran-Mantel-Haenszel — P-value derived from CMH General Association Test adjusting for region and weight group; Response ratio > 1 favors aripiprazole; Response ratio = 1.61, 95% CI 2-sided [1.20 to 2.16]

6. Secondary Outcome: Treatment Discontinuation Rate
Description: Treatment discontinuation rate will be calculated as the number of discontinued participants (ie, those who were withdrawn from the trial without completing the Week 8 visit) over the number of all randomized participants.
Time Frame: Week 8
Population: ITT Population: All participants randomly assigned to the double-blind treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Aripiprazole Low Dose | Aripiprazole High Dose | Placebo
Number analyzed (Participants) | 44 | 45 | 44
Percentage of participants | 4.5 | 22.5 | 4.5
Statistical Analysis 1: Comparison: Aripiprazole Low Dose vs Placebo; Test type: Superiority or Other; p = 0.9187, Cochran-Mantel-Haenszel — Discontinuation ratio < 1 favors aripiprazole. P-value derived from CMH General Association Test adjusting for region and weight group; Discontinuation ratio = 1.16, 95% CI 2-sided [0.19 to 7.05]
Statistical Analysis 2: Comparison: Aripiprazole Low Dose vs Placebo; Test type: Superiority or Other; p = 0.9576, Regression, Cox — Hazard ratio < 1 favors aripiprazole. P-value derived from Cox proportional hazard regression adjusting for region and weight group; Hazard Ratio (HR) = 1.05
Statistical Analysis 3: Comparison: Aripiprazole High Dose vs Placebo; Test type: Superiority or Other; p = 0.0132, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]; Discontinuation ratio = 4.06, 95% CI 2-sided [1.10 to 14.95]
Statistical Analysis 4: Comparison: Aripiprazole High Dose vs Placebo; Test type: Superiority or Other; p = 0.0278, Regression, Cox — [p-value comment as in outcome 6, analysis 2]; Hazard Ratio (HR) = 5.51

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the time of signing the informed consent up to 30 days after the last trial visit.
Description: An AE is defined as any untoward medical occurrence with the use of study drug. AE was considered serious if fatal, life threatening, disabling or incapacitating, required in participant hospitalization or prolonged hospitalization, congenital anomaly/birth defect or other medically significant event.
Arm/Group | Aripiprazole Low Dose | Aripiprazole High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 21/44 | 29/45 | 8/44
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole Low Dose (N=44) | Aripiprazole High Dose (N=45) | Placebo (N=44)
Nausea (Gastrointestinal disorders) | 3 | 4 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 2
Fatigue (General disorders) | 3 | 7 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4 | 0
Increased appetite (Metabolism and nutrition disorders) | 4 | 3 | 1
Akathisia (Nervous system disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 3 | 4 | 1
Lethargy (Nervous system disorders) | 0 | 5 | 0
Sedation (Nervous system disorders) | 8 | 4 | 1
Somnolence (Nervous system disorders) | 5 | 7 | 1
Restlessness (Psychiatric disorders) | 0 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No